CLINICAL TRIAL: NCT03877653
Title: Double-Blinded Randomized Control Trial of Knee Pain Utilizing Sub-Threshold Peripheral Nerve Stimulation
Brief Title: Freedom-1 Study for Chronic Knee Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Collaborators: Texas Institute for Pain and spine (Unknown); Performance Pain and Sports Medicine PLLC (Unknown); Holy Cross Hospital, Inc (Unknown); Colorado pain Care, LLC (Unknown); Advanced Spine and Pain (Unknown); Desert Orthopaedic Institute (Unknown); Vista Clinical Research (Unknown); Premier Pain Treatment (Unknown); Florida Joint Pain Institute (Unknown); Austin Orthopedic Institute (Unknown); Kettering Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30-00946; Freedom-1 (Other: Curonix)
Record Dates: First submitted 2019-02-11; First posted 2019-03-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritic Knee Pain
Keywords: PNS; Chronic; Pain; Wireless; Neuromodulation; knee; osteoarthritic; peripheral nerve stimulation; infra patellar saphenous
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: placebo-controlled double blinded randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A sponsor representative will open the sealed envelopes and assign groups. Investigators and research staff will be blinded to assignment of high frequency or sham. Randomization assignment will be documented post-implant but will be filed separately in a document locker, which will only be available to a sponsor representative until the time of unblinding.
  When receiving active stimulation, devices will be programmed to deliver electrical stimulation below perception threshold. Stimulation waveforms delivered above perception threshold have the potential to unblind subjects to their assignments.
  When receiving sham stimulation, devices will be programmed to not actively deliver electrical stimulation but still deplete battery life to maintain blinding. Subjects will have to recharge batteries similar to receiving active stimulation.
  Sites will not have access to the programmer. Study devices can only be programmed by Stimwave representatives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional (Experimental): Single arm, active stimulation
  Interventions: Device: Wireless neuromodulation
- Placebo (Placebo Comparator): When receiving sham stimulation, devices will be programmed to not actively deliver electrical stimulation but still deplete battery life to maintain blinding. Subjects will have to recharge batteries similar to receiving active stimulation.
  Sites will not have access to WaveCrest programmer. Study devices can only be programmed by Stimwave representatives.
  Interventions: Device: Wireless neuromodulation

INTERVENTIONS:
Device: Wireless neuromodulation — A needle and catheter are carefully inserted near the enervated nerve. The stimulator is then placed through the catheter close to the nerve. The proximal end of the stimulator is then sutured underneath the skin to prevent migration.

SUMMARY:
To demonstrate the potential benefits and risk of active sub-threshold stimulation in the treatment of chronic knee pain as compared to subjects that did not have active stimulation. Improvement will be assessed in relation to the clinical outcome measures of pain, with primary endpoint; Pain relief rate as measured by the number of subjects with greater or equal to a 50% decrease in pain on the visual analog scale, comparing baseline to the 1-month follow-up.

DETAILED DESCRIPTION:
Screening and Patient Selection Subjects will be selected from the pool patients of routine care who meet all the inclusion criteria for this study and none of the exclusion criteria, as described in Section 9.3.

Candidates will be given a patient information sheet (or Informed Consent) either in clinic or sent via post. Each approached candidate will be logged, assigned a screening number, and evaluated by the site research team. Subjects who sign the Informed Consent for participation and meet the Inclusion and Exclusion criteria will be enrolled and listed with an enrollment number. Recruitment will continue competitively until at least 84 subjects have evaluable data for evaluation of the primary endpoint.

Average pain levels will be captured at screening/baseline. Diagnostic Injection A diagnostic injection of the IPS under ultrasound, fluoroscopy or landmark guided in the clinic will be performed administering no more than 2cc of anesthetic. No steroids are allowed for the diagnostic injection. Only those subjects with significant temporary pain relief (> 75%) compared to the average pain level captured at baseline, and after at least 2 hours of the injection, will be allowed to continue with the study.

Trial Implant All subjects will be brought to the procedure room or operating room (OR) for the trial implant procedure under local anesthetic. An introducer will be placed under ultrasound or fluoroscopic guidance at the target nerve and the electrodes percutaneously advanced towards the IPS. After insertion of the receiver and then confirmation of stimulation, the trial stimulator will be secured to the skin. The stimulator tail will be outside the body and attached to the skin. All subjects will undergo an active 7-day provisional test period. Only those subjects reporting > 50% pain relief at the end of the 7-day provisional test period as compared to the average pain level captured at baseline will be allowed to continue with the study. The trial leads will be removed at the end of 7 days.

Permanent Implant All subjects responding to therapy with > 50% pain relief at 7 days will, at a later date, be brought to the operating room (OR) and given a sedative and local anesthetic for implantation of a permanent electrode. An introducer will be placed under ultrasound or fluoroscopic guidance onto the target nerve and the electrode array advanced towards the nerve. The receiver will be mated with the electrode array, and, after confirmation of stimulation, the permanent stimulator will be tunneled and secured. The device will remain inactive for 10 days to allow for satisfactory healing. If no localized infection or other complication, subjects can be brought back to the office for randomization.

Randomization/Blinding Subjects will be randomized to either active sub-threshold (high frequency) stimulation or no stimulation (sham) by Curonix's Clinical Support. All subjects, the investigator and the research team will be blinded to the group assignment for up to 30 days from the moment of randomization.

Office Study Visits After randomization follow-up visits will be conducted at 1 week, 1 month, 3 months, and 6 months.

Initial and follow-up evaluations will consist of physical exams, pain scale (m-MPS), Knee Injury & Osteoarthritis Outcome Score Junior (KOOS Jr), range of motion (flexion and extension measured by goniometer, work status and medication intake evaluation. At 1-month post-randomization, all subjects will be unblinded. Active devices can be adjusted for optimal pain relief. Sham devices will be reprogrammed to receive active treatment.

Available stimulation programs include tonic (on table testing), 500 Hz, 1000 Hz 1499 Hz frequency stimulation, all of which may be utilized on the same subject.

Remote Study Visits Follow up phone calls at 12 months, 18 months, and 24 months post-implantation will be performed to confirm durability of pain relief with the m-MPS and the global perceived effects scale (GPES). Any adverse events will be assessed and captured as part of the study.

ELIGIBILITY:
Inclusion Criteria:

i. Subject is over 18 years of age; ii. Subjects with a history of chronic, function-limiting (m-MPS >6/10) knee pain from osteoarthritis of at least three months in duration with or without prior surgeries; iii. Subject has been diagnosed with Kellgren-Lawrence Grade II or III knee osteoarthritis, confirmed by X-ray studies conducted in the last year; iv. Subject has been examined and has been deemed to be an appropriate candidate for the procedure, including chronic knee pain in patients post total knee replacement (TKR); v. Subjects who are able to understand this investigation, and give voluntary, written informed consent to participate in this study; vi. Subjects who are able to co-operate with the study procedures and are willing to return to the center for all the required post-operative follow-ups; vii. Documented failure of at least two less invasive treatment modalities including physical therapy, intra-articular steroids and/or oral NSAIDS; viii. Subject has not had recent invasive surgical procedures of the knee within the following intervals in relation to the time of signing Informed Consent:- 2 weeks for steroid injection - 4 weeks for radiofrequency, cryoablation or hyaluronic acid (HA) injection ix. Subject noted good (> 75%) but only temporary relief for at least 2 hours from an infrapatellar saphenous nerve injection with local anesthetic; x. Subject is deemed to be neuro-psycho-socially appropriate for implantation therapies based of assessment of a Clinical Psychologist.

Exclusion Criteria:

xi. Significant contralateral knee pain that would influence their level of activity greater to 6 on the modified-Mankosky Pain Scale; xii. Hip or foot pain greater than knee pain; xiii. Neurogenic or vascular claudication; xiv. Subject has been diagnosed with Kellgren-Lawrence Grade IV knee osteoarthritis, confirmed by X-ray studies conducted in the last year; xv. Uncontrolled major depression or uncontrolled psychiatric disorders; xvi. Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, infection, unstable angina, and severe chronic obstructive pulmonary disease; xvii. Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function (eg. Rheumatoid arthritis, severe spinal stenosis, activity-limiting cardiac disease); xviii. Women who are pregnant or planning to become pregnant, lactating; xix. Body mass index (BMI) greater than 40 (morbid obesity); xx. Subjects with multiple complaints involving concomitant knee, foot, or ankle pathology or radiculopathy, that will not be amenable to study due to the overlap of pain complaints; xxi. Subject has been examined and has been deemed to be inappropriate for the procedure based on anatomical restrictions; xxii. Lymphedema or stasis ulcers or other conditions that would compromise the surgical site; xxiii. History of adverse reaction to local anesthetic drugs; xxiv. Worker's compensation claimants; xxv. Incarcerated or has an ankle position locator; xxvi. Documented allergy to device material components; xxvii. Known or suspected substance abuse within the last 2 years; xxviii. Pacemaker or implanted defibrillator; xxix. Participation in another clinical study that could confound the results of this study; xxx. Based on the opinion of the investigator any legal or medical concerns that would preclude his/her enrollment in the study or potentially confound the results; xxxi. Any other implanted active medical devices in the same site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Responder rate | 1 month
  A. Percentage of patients with at least 50% improvement in the knee pain identified at baseline compared to 3 months post full implant of the StimQ PNS System pain identified at baseline compared to 6 months post full implant of the Freedom PNS system with the VAS

SECONDARY OUTCOMES:
Mankoski pain scale | 1 month
  The Mankoski Pain Scale is a numerical scale from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable. As pain is a subjective experience and individuals may interpret the severity of their pain differently, the MPS includes descriptions of each level of pain intensity to standardize the pain interpretation across subjects enrolled in this study.
Koos Jr | 1 month
  The KOOS assesses patient knee pain, function in daily living, function in sport and recreation, and knee related quality of life. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, useful for assessing changes in knee pathology over time, with or without treatment
Global Perceived Effect scales (GPES) | 1 month
  Patient satisfaction with the implant will be measured by assessing global perceived effects (GPES) on a 7-point scale (1 = worst and 7 = best) Scale from 1 (no change) to 7 (a great deal better) describing improvement with therapy
McGill Short Form (SF-MPQ-2) | 1 month
  The SF-MPQ-2 is a patient self-reported depression and pain quality questionnaire consisting of 22 questions, with all questions scored on a scale of 0 to 10. Answers on a scale of 0 (none) to 10 (worst possible)
Neuropathic pain questionnaire (DN4) | baseline
  The DN4 is a patient self-reported questionnaire designed to evaluate to degree of neuropathic pain. There are 10 questions on a scale of 0 (No) to 1 (Yes). Scores equal or higher than 4 out of 10 are an indication for the presence of neuropathic pain.
Work status (if working); | 1 month
  Work history and status will be evaluated based on a patient's self-reported questionnaire(s) completed at screening/baseline and all follow up visits.
Percentage Increase in Ability to do Knee Bends and Walking Tolerance | 1 month
  The patients will be evaluated for knee bends and walking tolerance before and after the treatment, using a treadmill for distance. Scale in degrees and (k)meters
Range of Motion | 1 month
  The passive and active range of motion will be measures with a goniometer.
Timed Up & Go (TUG) | 1 month
  This test assesses mobility. The patient sits back in a standard armchair, and identifies a line on the floor 3 meters (10 feet) away. When the examiner says "go", the patient is timed to see how long it takes to get up out of the chair, walk to the line, turn around, come back to the chair and sit down
Medication: Change in concomitant pain medication usage | 1 month
  Measure a change in concomitant pain medication usage.

OTHER OUTCOMES:
Treadmill | 1 month
  Pain-free walking time and distance on the treadmill

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Western Clinical Research, Placentia, California
  - Colorado Pain Care, LLC, Denver, Colorado
  - Holy Cross Hospital, Inc, Fort Lauderdale, Florida
  - Florida Joint Care Institute, Trinity, Florida
  - Southern Pain and research, Jasper, Georgia
  - Vista Clinical Research/Summit Spine & Joint Centers, Newnan, Georgia
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - Orthopedic Associates of Southwest Ohio, Dayton, Ohio
  - Premier Pain Treatment, Loveland, Ohio
  - Kettering Health, Miamisburg, Ohio
  - Austin Orthopedic Institute, Austin, Texas
  - Performance pain and sports medicine, Houston, Texas
  - Advanced Spine and Pain Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No